CLINICAL TRIAL: NCT04971564
Title: Thrombo-inflammation Biomarkers Trial in Acute Cerebral Hypoxia. A Case-control Trial Nested in a Cohort
Brief Title: Thrombo-inflammation Biomarkers Trial in Acute Cerebral Hypoxia
Acronym: RADICAL
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: FDE_2021_19
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Hypoxia; Ischemic Stroke
MeSH Terms: conditions — Hypoxia, Brain; Ischemic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with cerebral hypoxia victims of ischaemic stroke, acute parenchymal haemorrhage or subarachnoid haemorrhage
  Interventions: Other: Blood sampling
- Control: Patients without cerebral hypoxia
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling will be made to Day 0, Day 3 and to 3 month after inclusion

SUMMARY:
The goal of this trial is to study, in three well-defined clinical situations responsible for cerebral hypoxia, the concentrations of biomarkers of thrombo-inflammation compared to a population of patients without cerebral hypoxia, and to study in patients with cerebral hypoxia the association between these concentrations and the clinical evolution.

ELIGIBILITY:
Inclusion Criteria:

- For cases, admitted within the first 36 hours of an acute neurological symptom related to :

* An ischaemic cerebrovascular accident (iCVA) eligible for a mechanical thrombectomy procedure,
* A subarachnoid haemorrhage (SAH, all aetiologies) : patient presenting with at least a modified Fisher scale 3 or 4,
* An intra-parenchymal haematoma (IPH) with greatest axis ≥ 20mm or with NIHSS on admission >4.

OR

* For control patients, admitted within 7 days of the onset of acute neurological symptomatology related to a clinical diagnosis of transient ischaemic attack (TIA) - based on thorough questioning of the patient on admission - and prior to imaging, with an ABCD2≥ 2 score.
* Express consent to participate in the study.
* Member or beneficiary of a social security.

Exclusion Criteria:

* Pre-existing functional and/or cognitive disability
* Patient under legal protection.
* Pregnant or breastfeeding woman.
* Patient with secondary haemorrhagic transformation.

Secondary exclusion criteria :

* Patients with an ischaemic lesion visible on imaging, unrelated to large vessel occlusion and therefore ineligible for mechanical thrombectomy.
* Patients diagnosed with an acute non-vascular neurological pathology (migraine, epilepsy, etc.).
* TIA patients presenting an abnormality on follow-up imaging 24-48 hours after the initial imaging.

Excluded patients will be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Rothschild Foundation Hospital within the first 24 hours of an acute neurological symptomatology
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Biomarker rates at day 0 | 24 hours
  Biomarker: Neutro-Plaket aggregates, extra-cellular DNA networks, von Willebrand Factor

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France